CLINICAL TRIAL: NCT03444766
Title: Safety Study of Nivolumab for Selected Advanced Malignancies in India
Brief Title: Study of Nivolumab for Advanced Cancers in India
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-887
Record Dates: First submitted 2018-02-20; First posted 2018-02-23 (Actual); Results first posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC); Non-Small-Cell Lung Carcinoma; Nonsmall Cell Lung Cancer; Kidney Cancer; Kidney Neoplasms; Renal Cancer; Renal Neoplasms
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Kidney Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Monotherapy (Experimental): administering nivolumab only
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — specified dose on specified days
  Other Names: Opdivo

SUMMARY:
This is a study of nivolumab in participants with advanced Non-Small Cell Lung Cancer or Kidney Cancer in India.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Locally advanced or metastatic non-small cell lung cancer (NSCLC) after prior chemotherapy OR advanced renal cell carcinoma (RCC) after prior therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1
* Prior radiotherapy or radiosurgery must have been completed at least 2 weeks prior to randomization

Exclusion Criteria:

* Participants with untreated, symptomatic central nervous system (CNS) metastases
* Participants with carcinomatous meningitis
* Participants with active, known or suspected autoimmune disease
* Participants with a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications
* Other active malignancy requiring concurrent intervention

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (8):
- India (8):
  - Local Institution, Bangalore
  - Local Institution, Bengaluru
  - Local Institution, Hyderabad
  - Local Institution, Jaipur
  - Local Institution, Kolkata
  - Local Institution, Mumbai
  - Local Institution, New Delhi
  - Local Institution, Vellore

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 100 participants treated
Groups:
- Nivolumab: 3mg/kg IV q 2weeks
Period: Overall Study
Arm/Group | Nivolumab
Started (Started Treatment Period) | 100
Completed (Completed Treatment Period) | 34
Not Completed | 66
Not completed — Other Reasons | 2
Not completed — Participant Withdrew Consent | 5
Not completed — Lost to Follow-up | 2
Not completed — Death | 2
Not completed — Adverse Event Unrelated to Study Drug | 6
Not completed — Disease Progression | 49

BASELINE CHARACTERISTICS:
Arm/Group | Nivolumab
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.7 (10.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 100
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 100
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events
Description: Number of participants with treatment-related Adverse Events based on worst ctc grade
  Includes events reported between first dose and 100 days after last dose of Nivolumab or for a total of 26 weeks from first on-study treatment with Nivolumab whichever is earliest.
Time Frame: 26 Weeks
Population: All treated participants
Measure: Number; unit: Count of participants
Arm/Group | Nivolumab
Number analyzed (Participants) | 100
Count of participants
  Any Grade | 25
  Grade 3-4 | 4
  Grade 5 | 1

2. Secondary Outcome: Number of Participants With Treatment-related Select Adverse Events
Description: Number of participants with treatment-related Select Adverse Events based on worst ctc grade for the following categories:
  Pulmonary, Gastrointestinal, Endocrinopathies, Hepatic, Renal, Skin, Neurological and Hypersensitivity/Infusion reactions
  Includes events reported between first dose and 100 days after last dose of Nivolumab or for a total of 26 weeks from first on-study treatment with Nivolumab whichever is earliest.
Time Frame: 26 Weeks
Population: All treated participants
Measure: Number; unit: Count of participants
Arm/Group | Nivolumab
Number analyzed (Participants) | 100
Count of participants
  Pulmonary (Grade 3) | 1
  Pulmonary (Grade 5) | 1
  Hepatic (Grade 1) | 1
  Skin (Grade 1) | 2
  Hypersensitivity/Infusion reaction (Grade 1) | 1
  Hypersensitivity/Infusion reaction (Grade 2) | 2

3. Secondary Outcome: Number of Participants With Treatment-related Serious Adverse Events
Description: Number of participants with treatment-related Serious Adverse Events based on worst CTC grade
  Includes events reported between first dose and 100 days after last dose of Nivolumab or for a total of 26 weeks from first on-study treatment with Nivolumab whichever is earliest.
Time Frame: 26 Weeks
Population: All treated participants
Measure: Number; unit: Count of participants
Arm/Group | Nivolumab
Number analyzed (Participants) | 100
Count of participants
  Any Grade | 4
  Grade 3 - 4 | 3
  Grade 5 | 1

4. Secondary Outcome: Number of Participants With Adverse Events Leading to Discontinuation
Description: Number of participants with Adverse events leading to discontinuation of treatment based on worst CTC grade
  Includes events reported between first dose and 100 days after last dose of Nivolumab or for a total of 26 weeks from first on-study treatment with Nivolumab whichever is earliest.
Time Frame: 26 Weeks
Population: All treated participants
Measure: Number; unit: Count of participants
Arm/Group | Nivolumab
Number analyzed (Participants) | 100
Count of participants
  Grade 1 | 7
  Grade 2 | 5
  Grade 3 | 9
  Grade 4 | 0
  Grade 5 | 1

ADVERSE EVENTS:
Time Frame: 26 Weeks
Description: Includes events reported between first dose and 100 days after last dose of Nivolumab or for a total of 26 weeks from first on-study treatment with Nivolumab whichever is earliest.
Arm/Group | Nivolumab
All-Cause Mortality (participants affected / at risk) | 17/100
Serious Adverse Events (participants affected / at risk) | 30/100
Other Adverse Events (participants affected / at risk) | 74/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab (N=100)
Cardiac arrest (Cardiac disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 3
Pyrexia (General disorders) | 1
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Malaria (Infections and infestations) | 1
Respiratory tract infection viral (Infections and infestations) | 1
Blood electrolytes abnormal (Investigations) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Pseudohyperkalaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab (N=100)
Anaemia (Blood and lymphatic system disorders) | 8
Hypothyroidism (Endocrine disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 10
Diarrhoea (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 17
Asthenia (General disorders) | 6
Chest pain (General disorders) | 11
Fatigue (General disorders) | 16
Pyrexia (General disorders) | 21
Decreased appetite (Metabolism and nutrition disorders) | 11
Hyponatraemia (Metabolism and nutrition disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 13
Headache (Nervous system disorders) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 24
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-05-07): https://cdn.clinicaltrials.gov/large-docs/66/NCT03444766/SAP_000.pdf
  • Study Protocol (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT03444766/Prot_001.pdf